CLINICAL TRIAL: NCT04573738
Title: Safety and Feasibility Study of Robotic Assisted Transanal Total Mesorectal Excision for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Professor, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200913
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer; Perioperative Complication
Keywords: Rectal Cancer; Robotic surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic transanal surgery (Experimental): Robotic assisted transanal total mesorectal excision for rectal cancer patients
  Interventions: Procedure: Robotic assisted transanal total mesorectal excision
- Laparoscopic transanal surgery (Active Comparator): Laparoscopic transanal total mesorectal excision for rectal cancer patients
  Interventions: Procedure: Laparoscopic assisted transanal total mesorectal excision

INTERVENTIONS:
Procedure: Robotic assisted transanal total mesorectal excision — Robotic assisted transanal total mesorectal excision for rectal cancer patients
  Arms: Robotic transanal surgery
Procedure: Laparoscopic assisted transanal total mesorectal excision — Laparoscopic assisted transanal total mesorectal excision for rectal cancer patients
  Arms: Laparoscopic transanal surgery

SUMMARY:
Total mesorectal excision has greatly reduced the local recurrence rate of rectal cancer after colorectal surgery. Transanal total mesorectal excision(TaTME) is potentially a suitable option for patients with middle and low rectal cancer. Robotic systems are expected to develop the advantages of TaTME to overcome the limitations of laparoscopic surgery. This study aimed to investigate the safety and feasibility of robotic assisted transanal total mesorectal excision in patients with rectal cancer.

DETAILED DESCRIPTION:
TaTME is potentially a suitable option for patients with middle or low rectal cancer, especially for males with obesity and a narrow pelvis.The da Vinci robotic system (Intuitive Surgical, Sunnyvale, CA, USA) is expected to overcome the limitations of the laparoscopic transanal approach for rectal surgery. Da Vinci Si Surgical System or da Vinci Xi Surgical System would be used to performed Transanal total mesorectal excision. And the surgery would performed by two-team approach. This study aimed to investigate the safety and feasibility of robotic assisted transanal total mesorectal excision in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological biopsy confirmed adenocarcinoma of the rectum.
2. Preoperative assessment of tolerance to surgery without major organ dysfunction.
3. Patients must be able to understand and voluntarily sign written informed consent.
4. The surgical method is robotic assisted transanal total mesorectal excision
5. Distance of the edge of the tumour within 8 cm

Exclusion Criteria:

1. The patient cannot tolerate the operation.
2. Refusal to sign informed consent.
3. Patients with distant metastasis of rectal cancer.
4. The surgical method was changed to miles or Hartman;
5. Unable to complete the follow - up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The local recurrence rates of rectal cancer | Two years after surgery
  The incidence of local recurrence rectal cancer within two years after surgery
The incidence of postoperative anastomotic leakage | Within 30 days after surgery
  The incidence of postoperative anastomotic leakage within 30 days after surgery
The five-year survival rates | Five years after surgery
  The 5-year survival rates of rectal cancer
The distant metastasis rates of rectal cancer | Five years after surgery
  The incidence of distant metastasis rectal cancer within two years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, MD, Study Chair — Army Military Medical University
Locations (1):
- Daping hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee L, de Lacy B, Gomez Ruiz M, Liberman AS, Albert MR, Monson JRT, Lacy A, Kim SH, Atallah SB. A Multicenter Matched Comparison of Transanal and Robotic Total Mesorectal Excision for Mid and Low-rectal Adenocarcinoma. Ann Surg. 2019 Dec;270(6):1110-1116. doi: 10.1097/SLA.0000000000002862. PMID 29916871
- [Background] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Background] Atallah S, Martin-Perez B, Pinan J, Quinteros F, Schoonyoung H, Albert M, Larach S. Robotic transanal total mesorectal excision: a pilot study. Tech Coloproctol. 2014 Nov;18(11):1047-53. doi: 10.1007/s10151-014-1181-5. Epub 2014 Jun 24. PMID 24957360
- [Background] Ye J, Tian Y, Wang L, Ye Y, Zhang Y, Li F, Liu B, Tong W. [Robotic-assisted transanal total mesorectal excision for lower rectal cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2017 Aug 25;20(8):900-903. Chinese. PMID 28836251